CLINICAL TRIAL: NCT01160484
Title: A Phase II Study of Pegylated Liposomal Doxorubicin, Bortezomib, Dexamethasone and Lenalidomide (DVD-R) for Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Pegylated Liposomal Doxorubicin, Bortezomib, Dexamethasone and Lenalidomide for Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncotherapeutics (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-MM-PI-0533
Record Dates: First submitted 2010-07-07; First posted 2010-07-12 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; refractory; relapsed; bortezomib; doxil
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Calcium Dobesilate; Bortezomib; liposomal doxorubicin; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVD-R single arm (Experimental): Dose schematic of Dexamethasone + Bortezomib + Pegylated Liposomal Doxorubicin + Lenalidomide (DVD-R) Therapy:
  Dexamethasone*- 40 mg IV Bortezomib**- 1.0 mg/m2 IV Push Pegylated Liposomal Doxorubicin*- 4.0 mg/m2 IV Lenalidomide***- 10 mg PO
  Per 28 Day Cycle
  * Intravenous infusion (IV) Days 1, 4, 8 and 11 ** Intravenous push (IVP) Days 1, 4, 8 and 11 *** Per Orem (PO) Days 1-14
  Interventions: Drug: DVD-R

INTERVENTIONS:
Drug: DVD-R — 40 mg dexamethasone will be administered IV on Days 1, 4, 8, and 11 of each cycle. 1.0 mg/m2 Bortezomib will be administered IV over 3 to 5 seconds followed by a standard saline flush, on Days 1, 4, 8, and 11 immediately following the dexamethasone infusion. 4.0 mg/m2 PLD will be given as a 90 minute infusion on Day 1 of Cycle 1 and subsequent doses may be administered over 30 to 60 minutes on Days 4, 8 and 11 of Cycle 1 and on Days 1, 4, 8, and 11 of each subsequent cycle, following the bortezomib administration. 10 mg/day lenalidomide will be administered PO on days 1-14 of a 28-day treatment cycle, followed by a 14-day rest period, following the PLD administration.
  Other Names: Decadron, Velcade, Doxil, Revlimid

SUMMARY:
This is a phase II, multicenter, open label, nonrandomized study to evaluate the efficacy and safety of lenalidomide at a dose of 10 mg/dose in combination with bortezomib at 1.0 mg/m2/dose, pegylated liposomal doxorubicin (PLD) at 4.0 mg/m2/dose, and intravenous (IV) dexamethasone at 40 mg/dose in adult patients with relapsed/refractory multiple myeloma (MM). The study consists of a screening period, followed by up to eight 28 day open label treatment cycles, a final assessment to occur 28 days after the end of the last treatment cycle, and a follow-up period.

DETAILED DESCRIPTION:
Studies have shown that combinations of PLD and bortezomib have striking synergy in preclinical studies and impressive response rates (73 & 89%) in early clinical trials for MM patients with relapsed/refractory disease as well as first-line therapy. In addition, the efficacy of PLD with bortezomib in anthracycline-insensitive patients has been greater than single-agent bortezomib when comparing across studies. The immunomodulatory drugs, thalidomide and lenalidomide, target the tumor cell microenvironment, are antiangiogenic, have an immune activation effect and also exert a direct cytotoxic effect on myeloma cells. A phase 1 clinical study by our group also demonstrated that low dose PLD, administered at a more frequent dosing schedule, in combination with bortezomib, and dexamethasone (DVD regimen) is well tolerated and associated with high response rates and durable responses. In this phase II prospective trial, we will evaluate this regimen and show that this change enhances the DVD-R regimen's safety and efficacy for patients with relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of multiple myeloma (MM) based on standard criteria (Durie 1986)
2. Currently has MM with measurable disease (serum m protein > 1.0g/dl and/or 24 hr urine m protein > 200mg/24 hr)
3. Currently has progressive MM that has relapsed or is refractory
4. Voluntarily signed an informed consent
5. Age 18 years
6. Eastern Cooperative Oncology Group (ECOG) performance < 2
7. Life-expectancy > 3 months
8. Laboratory test results within these ranges:

   * Absolute neutrophil count (ANC) 1.5 x 109/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then 1.0 x 109/L
   * Platelet count 75 x 109/L; if the bone marrow is extensively infiltrated (> 70% plasma cells) then 50 x 109/L
   * Hg > 8 g/dL
   * Calculated or measured creatinine clearance > 30 mL/minute.
   * Total bilirubin 2.0 x upper limit of normal (ULN)
   * Aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/serum glutamic pyruvic transaminase (ALT/SGPT) 3 x ULN or 5 x ULN if hepatic metastases are present
   * Serum potassium within the normal range
9. Disease free of prior malignancies for 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast
10. Registered into the mandatory RevAssist® program, willing and able to comply with the requirements of RevAssist®.
11. Females of childbearing potential must have a negative serum or urine pregnancy test and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control.
12. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin)

Exclusion Criteria:

1. Plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes syndrome
2. Plasma cell leukemia
3. Grade 2 peripheral neuropathy within 14 days before enrollment
4. Impaired cardiac function or clinically significant cardiac diseases, including myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class II or greater heart failure, Uncontrolled angina, clinically significant pericardial disease, severe uncontrolled ventricular arrhythmias, echocardiogram or Multigated acquisition(MUGA) scan evidence of left ventricular ejection fraction (LVEF) below institutional normal within 28 days prior to enrollment, electrocardiographic (ECG) evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
5. Severe hypercalcemia, i.e., serum calcium 12 mg/dL (3.0 mmol/L) corrected for albumin
6. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
7. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
8. Undergone major surgery within 28 days prior enrollment or has not recovered from side effects of such therapy (Kyphoplasty is not considered to be a major surgery; however, the investigator is to discuss enrollment of a patient with a recent history of kyphoplasty with the medical monitor).
9. Pregnant or breast feeding females. (Lactating females must agree not to breast feed while taking lenalidomide)
10. Received the following prior therapy:

    * Chemotherapy within 3 weeks of enrollment (6 wks for nitrosoureas)
    * Corticosteroids (>10 mg/day prednisone or equivalent) within 3 weeks of enrollment
    * Immunotherapy or antibody therapy as well as thalidomide, lenalidomide, arsenic trioxide or bortezomib within 21 days before enrollment
    * Radiation therapy within 28 days before enrollment, except localized radiation therapy
    * Use of any other experimental drug or therapy within 28 days of enrollment
11. Known hypersensitivity to compounds of similar to thalidomide, doxorubicin, bortezomib, boron or mannitol.
12. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
13. Concurrent use of other anti-cancer agents or treatments
14. Known positivity for human immunodeficiency virus (HIV) or hepatitis B or C; baseline testing for HIV and hepatitis B or C is not required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R. Berenson, MD, Principal Investigator — James R. Berenson, MD, Inc.
Locations (8):
- United States (8):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Hematology-Oncology Medical Group of Fresno, Inc., Fresno, California
  - Loma Linda University, Loma Linda, California
  - Santa Barbara Hematology Oncology, Santa Barbara, California
  - James R. Berenson, M.D., Inc., West Hollywood, California
  - Watson Clinic, LLP, Center for Care and Research, Lakeland, Florida
  - Bassett Cancer Institute, Cooperstown, New York
  - Broome Oncology, Johnson City, New York

REFERENCES:
- [Result] Berenson JR, Yellin O, Kazamel T, Hilger JD, Chen CS, Cartmell A, Woliver T, Flam M, Bravin E, Nassir Y, Vescio R, Swift RA. A phase 2 study of pegylated liposomal doxorubicin, bortezomib, dexamethasone and lenalidomide for patients with relapsed/refractory multiple myeloma. Leukemia. 2012 Jul;26(7):1675-80. doi: 10.1038/leu.2012.51. Epub 2012 Feb 22. PMID 22354206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from eight different clinical sites sites in the United States. Data was collected from September 2009 until July 25, 2011
Groups:
- DVD-R Single Arm: Dose schematic of Dexamethasone + Bortezomib + Pegylated Liposomal Doxorubicin (PLD)+ Lenalidomide (DVD-R) Therapy:
  Per 28 Day Cycle, patients will received drug in the following order, dosing and schedule:
  1) Dexamethasone- 40 mg intravenous infusion (IV) on Days 1, 4, 8 and 11; 2) Bortezomib- 1.0 mg/m2 infused over 3 to 5 seconds followed by a standard saline flush on Days 1, 4, 8 and 11; 3) Pegylated Liposomal Doxorubicin- 4.0 mg/m2 IV as a 90 minute infusion on Day 1 of Cycle 1 and subsequent doses may be administered over 30 to 60 minutes on Days 4, 8 and 11 of Cycle 1 and on Days 1, 4, 8, and 11 of each subsequent cycle; and 4) Lenalidomide- 10 mg PO on days 1-14
Period: Overall Study
Arm/Group | DVD-R Single Arm
Started | 40
Completed | 22
Not Completed | 18
Not completed — Lack of Efficacy | 9
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — inclusion/exclusion criteria failure | 1

BASELINE CHARACTERISTICS:
Population: The estimated number of participants will allow to determine whether the true rate of response to DVD-R is at least 50%, at the one-sided alpha-level of 0.05 and having at least 85% power
Groups:
- DVD-R Single Arm: Dose schematic of Dexamethasone + Bortezomib + Pegylated Liposomal Doxorubicin + Lenalidomide (DVD-R) Therapy:
  Per 28 Day Cycle, patients will received drug in the following order, dosing and schedule:
  1) Dexamethasone- 40 mg intravenous infusion (IV) on Days 1, 4, 8 and 11; 2) Bortezomib- 1.0 mg/m2 infused over 3 to 5 seconds followed by a standard saline flush on Days 1, 4, 8 and 11; 3) Pegylated Liposomal Doxorubicin- 4.0 mg/m2 IV as a 90 minute infusion on Day 1 of Cycle 1 and subsequent doses may be administered over 30 to 60 minutes on Days 4, 8 and 11 of Cycle 1 and on Days 1, 4, 8, and 11 of each subsequent cycle; and 4) Lenalidomide- 10 mg PO on days 1-14
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 27
Age, Continuous [Median (Full Range); unit: years] | 71 [34 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
International Staging System (ISS); stage (N) [Number; unit: participants]
  I (beta 2 microglobulin(B2M )<3.5 +Albumin ≥3.5) | 16
  II (B2M 3.5 +albumin < 3.5; or B2M 3.5-5.5) | 14
  III (B2M >5.5) | 10
Serum M-protein [Median (Full Range); unit: g/dL] | 2.05 [0.0 to 7.0]
Urine-M protein [Median (Full Range); unit: mg/dL] | 261.1 [0.0 to 7162.0]
Serum creatinine [Median (Full Range); unit: mg/dL] | 1.0 [0.6 to 3.4]
Prior treatments [Mean (Full Range); unit: number of treatments] | 3 [1 to 17]
Total Number of prior lines of treatment [Number; unit: number of treatments]
  Bortezomib (BTZ) | 33
  Alkylating agents | 20
  PLD or Doxorubucin | 15
  Thalidomide | 15
  Lenalidomide (LEN) | 19
  Glucocorticoids | 35
  HDAC inhibitors (panobinostat/romidepsin) | 7
  Transplant (autologous) | 5
  Other | 11
  PLD+btz+dexamethasone (dex) | 17
  PLD+btz+dex and len+ glucocorticoids | 10

OUTCOME MEASURES:

1. Primary Outcome: International Myeloma Working Group (IMWG) Response Criteria
Description: The investigator will evaluate each patient for response to therapy according to criteria augmented from those developed by Bladé et al., 1998 presented below (Table 7-1). Assessment of disease response will be performed prior to drug administration on Day 1 of Cycles 2 8 and at the End of Study Treatment visit. If a patient is determined to have complete response (CR), very good partial response (VGPR), partial response (PR), or minor response (MR), then assessment of disease response is to be performed 4 weeks later to confirm the response.
Time Frame: Up to 7.5 months (eight 28-day cycles)
Population: Population analysis was carried out as per protocol. Efficacy was evaluated via a modified version of the Bladé response criteria [complete response (CR), very good partial response (VGPR), partial response (PR), and those achieving minimal response (MR)]
Measure: Number; unit: participants
Groups:
- DVD-R Single Arm: 40 mg dexamethasone will be administered IV on Days 1, 4, 8, and 11 of each cycle. 1.0 mg/m2 Bortezomib will be administered IV over 3 to 5 seconds followed by a standard saline flush, on Days 1, 4, 8, and 11 immediately following the dexamethasone infusion. 4.0 mg/m2 PLD will be given as a 90 minute infusion on Day 1 of Cycle 1 and subsequent doses may be administered over 30 to 60 minutes on Days 4, 8 and 11 of Cycle 1 and on Days 1, 4, 8, and 11 of each subsequent cycle, following the bortezomib administration. 10 mg/day lenalidomide will be administered PO on days 1-14 of a 28-day treatment cycle, followed by a 14-day rest period, following the PLD administration.
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 39
participants
  CR | 8
  VGPR | 4
  PR | 7
  Objective Response (CR+VGPR+PR) | 19
  MR | 14
  Clinical Benefit (CR+VGPR+PR+MR) | 33
  Estable disease | 4
  Progressive disease | 2

2. Secondary Outcome: Time to First Response
Time Frame: Up to 7.5 months (eight 28-day cycles)
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 33
months | 1 [1 to 5]

3. Secondary Outcome: Time to Best Response
Time Frame: Up to 7.5 months (eight 28-day cycles)
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 33
months | 2 [1 to 6]

4. Secondary Outcome: Duration of Response
Time Frame: First evidence of PR or better (for overall response) and MR or better (for clinical benefit response) to start of disease progression or death.
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 33
months | 12 [1 to 21]

5. Secondary Outcome: Time to Progression
Time Frame: Time from the start of treatment to progressive disease
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 39
months | 9 [1 to 22]

6. Secondary Outcome: Progression-free Survival
Time Frame: Time from the start of treatment to progressive disease or until death
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 39
months | 9 [1 to 22]

7. Secondary Outcome: Follow-up Time
Description: time that patients were monitored for disease progression and overall survival
Time Frame: Follow-up visits for disease progression and overall survival every 3 months after study discontinuation. After progression, follow-up visits for survival status every 6 months or until alternate therapy needs to be started or death intervenes
Measure: Median (Full Range); unit: months
Arm/Group | DVD-R Single Arm
Number analyzed (Participants) | 39
months | 11 [2 to 22]

ADVERSE EVENTS:
Time Frame: Severity and frequency of adverse events (AEs) were evaluated at each visit. Serious adverse events (SAEs) were followed until resolution or until clearly determined be unrelated to study treatment.
Arm/Group | DVD-R Single Arm
Serious Adverse Events (participants affected / at risk) | 10/40
Other Adverse Events (participants affected / at risk) | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DVD-R Single Arm (N=40)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Disphagia (Gastrointestinal disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Loss of balance (General disorders) | 1 (1)
Pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic thrombophlebitis (Vascular disorders) | 1 (1)
Syncopal episode (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DVD-R Single Arm (N=40)
Fatigue (General disorders) | 16 (16)
Neutropenia (Blood and lymphatic system disorders) | 14 (14)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (14)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Edema (Blood and lymphatic system disorders) | 12 (12)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Periphenal neurophaty (Nervous system disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 10 (10)
Confusion (Psychiatric disorders) | 9 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 7 (7)
Pelvic pain (Reproductive system and breast disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Generalized pain (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No